CLINICAL TRIAL: NCT03551054
Title: Healthy for Two, Healthy for You: A Pilot Health Coaching Intervention for Pregnant Women
Brief Title: Healthy for Two, Healthy for You
Acronym: H42/H4U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Mid-Atlantic Nutrition Obesity Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00084709
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Weight Gain; Pregnancy Related
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy for Two, Healthy for You (Experimental): Remotely delivered behavioral health coaching in pregnancy and postpartum
  Interventions: Behavioral: Healthy for Two, Healthy for You
- Pregnancy Health Education (Active Comparator): Single health education visit with study staff member
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Healthy for Two, Healthy for You — Remotely delivered health coaching in pregnancy and postpartum to promote healthy weight gain.
  Arms: Healthy for Two, Healthy for You
Behavioral: Health Education
  Other Names: Single health education visit
  Arms: Pregnancy Health Education

SUMMARY:
Investigators conducted a pilot feasibility and acceptability randomized controlled trial of a remotely delivered behavioral health coaching program in pregnancy and postpartum.

DETAILED DESCRIPTION:
Half of pregnant women are overweight or obese. Obesity disproportionately impacts low-income women and women of racial and ethnic minorities. Maternal obesity is linked with adverse perinatal outcomes, including gestational diabetes and preeclampsia, as well as longer-term health problems such as obesity in offspring and maternal cardiovascular disease. Pregnancy provides a unique opportunity to engage women in improving their health behaviors because women are motivated to protect the health of their babies and have frequent interactions with the healthcare system. Advances in behavioral weight management and obesity prevention have not yet been translated into real-world prenatal care settings. Our team was recently supported by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)-funded Nutrition and Obesity Research Center Pilot and Feasibility program to adapt an evidence-based telephonic health coaching program for pregnant women. Investigators conducted 20 in-depth interviews with patients and providers to gain valuable feedback to inform the intervention design and delivery, and have put together a multi-disciplinary team to adapt the intervention. Investiagtors developed the intervention specific for pregnancy and postpartum based on this feedback and are testing the intervention, Healthy for Two / Healthy for You, to assess feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Mothers:

  * BMI >= 18.5 kg/m2 at time of eligibility screening
  * Age >=18
  * Able to provide informed consent
  * 12 weeks gestation or earlier
  * English speaking
  * Insurance type
  * Willing to provide address and >=2 contact people
  * Consistent use of a personal smartphone and willingness to use for health behavior tracking as part of the study
  * Patient at a participating prenatal clinical site
  * Access to internet (including public library and smartphone)
  * Demonstrated ability to track caloric intake for 4 days
  * Singleton pregnancy

Infants:

• Born during Mother's enrollment in study

Exclusion Criteria:

* • Type 1 or type 2 diabetes, pre-pregnancy or gestational diabetes, diagnosed prior to start of intervention (14 weeks gestation)

  * Multiple fetuses
  * Prior history of severe preeclampsia, pre-term birth (before 32 weeks gestation)
  * Prior history of or current diagnosis of incompetent cervix
  * Poorly controlled blood pressure (>160/100)
  * Unable to walk 1 block without pain, shortness of breath
  * Serious medication condition hindering use of recommendations for pregnancy weight gain
  * Not cleared by study's maternal-fetal medicine or treating obstetrician
  * Planning to relocate from areas in next 2 years
  * Psychiatric or substance use related hospitalization in past 1 year
  * (There is no exclusion criteria for the infants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy condition
Enrollment: 26 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | At 37 weeks gestation
  Gestational weight gain is calculated as weight, in pounds recorded at 37 weeks gestation minus the baseline weight recorded by 14 weeks gestation.

SECONDARY OUTCOMES:
Postpartum weight retention | At 3 months after delivery
  Postpartum weight retention is calculated as weight, in pounds, recorded at 3 months after delivery minus the weight recorded at baseline (by 14 weeks gestation).

IPD SHARING:
Plan to Share IPD: No